CLINICAL TRIAL: NCT06894966
Title: Targeted Therapeutic Transcranial Focused Ultrasound Intervention for Alcohol Use Disorder
Brief Title: Towards a Targeted Ultrasound Neuromodulation Intervention for Alcohol Abuse Disorders
Acronym: TUS-AUD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Elsa Fouragnan, Professor, University of Plymouth
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2024-4914-6227; MR/Y034368/1 (Other Grant/Funding Number: UKRI MRC)
Record Dates: First submitted 2025-02-27; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
Keywords: focused ultrasound; TUS; neuromodulation; AUD; Transcranial Ultrasound Stimulation
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Intervention Model Description: Within subject, randomized, double-blind, sham-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low intensity transcranial focused ultrasound stimulation (TUS) (Other): double-blind, sham-controlled, crossover study in N=30 individuals with OCD
  Interventions: Device: low intensity transcranial focused ultrasound stimulation (TUS)
- low intensity transcranial focused ultrasound stimulation (TUS) Sham (Other): double-blind, sham-controlled, crossover study in N=30 individuals with OCD
  Interventions: Device: low intensity transcranial focused ultrasound stimulation (TUS)

INTERVENTIONS:
Device: low intensity transcranial focused ultrasound stimulation (TUS) — Low-intensity transcranial focused ultrasound (TUS) provides an energy source with millimeter resolution that can be focused anywhere in the brain safely and effectively for non-invasive and transient neuromodulation. TUS is an important advance and of great significance for brain-mapping efforts, diagnostics, and therapies in neuroscience and particularly promising for addiction therapy as it provides unprecedented non-surgical access to the brain regardless of depth. Low intensities of focused ultrasound (TUS) are used so that tissue damage does not occur, but neural activity can be modulated by mechanical effects.

SUMMARY:
This study explores the potential of transcranial ultrasound stimulation (TUS) as an innovative therapeutic approach for individuals with Alcohol Use Disorder. By targeting specific brain regions associated with compulsive behaviors and reward dysfunction, the researchers aim to assess the safety and efficacy of TUS in reducing symptoms and enhancing cognitive flexibility.

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) is a prevalent and highly debilitating condition characterized by compulsive alcohol consumption, loss of control over drinking behavior, and significant impairment in social functioning and quality of life. Estimates suggest that the economic burden of AUD is substantial, with alcohol-related harm costing the UK over £21 billion per year (Public Health England, 2016). There is a pressing need for novel interventions that surpass current treatment approaches in both effectiveness and comprehensiveness, addressing the neural and behavioral mechanisms underlying AUD. Low-intensity transcranial focused ultrasound stimulation (TUS) is an emerging non-invasive brain stimulation technique with the potential to modulate neural activity with high spatial precision.

The neural basis of AUD involves dysfunction across several brain regions, including the prefrontal cortex (impaired executive control: Koob & Volkow, 2016), the striatum (habit formation and reinforcement: Everitt & Robbins, 2016), the amygdala (heightened stress reactivity: Koob, 2021), and the thalamus (altered sensory and reward processing: Müller-Oehring et al., 2015). TUS can precisely modulate neuronal activity in both cortical and subcortical regions, making it a promising tool for targeting the disrupted neurocircuitry of AUD. This study aims to explore the safety and efficacy of TUS in modulating key brain regions involved in compulsive alcohol use and cognitive control, with the goal of reducing AUD-related symptoms and improving treatment outcomes.

ELIGIBILITY:
Inclusion Criteria will be:

* Male or female, aged 21-55 years, and fluent English speaking.
* Participants score ≥ 20 on the AUDIT.
* Participant is willing and able to give informed consent for participation in the trial.
* Participant is willing to comply with all trial requirements and committed to participating in all six testing sessions.

Exclusion Criteria will be:

The participant may not enter the trial if ANY of the following apply.

History:

* serious head trauma or brain surgery
* (first-degree relatives with) epilepsy, convulsion, or seizure
* diagnosis of a neurological or psychiatric disorder (other than AUD)
* adverse reactions to non-invasive brain stimulation
* participation in another short-term non-invasive brain stimulation study in the past 3 days
* participation in another long-term non-invasive brain stimulation study in the past 28 days
* recent head trauma that was diagnosed as a concussion or associated with loss of consciousness

Current:

* pregnancy or planning a pregnancy during the course of the trial
* use of psychoactive drugs or any drugs listed in the Neurostimulation Safety Report
* heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement
* metal in the head or body
* claustrophobia
* extreme mood fluctuations
* predisposition to fainting spells (syncope)
* medication that will interfere with the study or constitutes an increased risk of adverse effects (e.g., affects brain excitability)
* hearing problems or ringing in the ears
* skin diseases or sensitivity at intended TUS stimulation site
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Last 24 hours:

* more than four alcoholic units
* recreational psychoactive drugs
* antibiotics

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2026-09-19 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Immediately after TUS session; one day and one week after TUS. Same for sham, to compare the TUS active and sham.
  number of adverse events

SECONDARY OUTCOMES:
Change in AUD symptoms | immediately prior to TUS sessions, within 1 hour post TUS and every day that follow TUS for 7 days
  numerical AUD symptoms rating scale and Alcohol Consumptions

CONTACTS AND LOCATIONS:
Locations (1):
- Health, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymous behavioral data upon publication
Supporting Information: SAP, Analytic Code
Time Frame: data will be available after analysis of primary and secondary outcomes are completed
Access Criteria: anyone with access to the link to the data (OSF)
URL: http://www.plymouth.ac.uk/students-and-family/governance/general-data-protection-regulation-gdpr

REFERENCES:
- See also: safety report for TUS use from expert consortium — https://arxiv.org/abs/2311.05359